CLINICAL TRIAL: NCT02655432
Title: Évaluation de l'Utilisation d'un Photoscreener Comme méthode de dépistage Des problèmes Ophtalmologiques pédiatriques en Haïti
Brief Title: Performance of a Photoscreener for Vision Screening in a Haitian Pediatric Population
Acronym: POPH
Status: Withdrawn | Type: Observational
Why Stopped: waiting for ethic board approval
Sponsor: Université de Montréal (Other)
Responsible Party: Principal Investigator, Patrick Hamel, Hospital chef of the ophthalmology department, CHU Sainte-Justine, Université de Montréal
Other Study IDs: 20160130
Record Dates: First submitted 2016-01-08; First posted 2016-01-14 (Estimated); Last update posted 2016-12-02 (Estimated); Status verified 2016-11

CONDITIONS: Amblyopia; Myopia; Hyperopia; Astigmatism; Cataract; Retinoblastoma; Trachoma; Xerophthalmia; Glaucoma; Retinopathy of Prematurity
MeSH Terms: conditions — Amblyopia; Myopia; Hyperopia; Astigmatism; Cataract; Retinoblastoma; Trachoma; Xerophthalmia; Glaucoma; Retinopathy of Prematurity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Spot photoscreener: Automated vision screener: Spot Vision Screener VS 100, Welch-Allyn. This photoscreener is a portable device, using an infrared light. It is built to detect amblyogenic risk factors. First of all, the spot photoscreener produces a sounds which attracts the child's attention and helps him shift his gaze towards the device, held at 1 meter in front him. The spot then evaluates for refractive errors, anisocoria, strabismus, ptosis and media opacity. The ophthalmologic evaluation consists of the measure of the visual acuity, ocular alignment, anterior and posterior segment. The patient will be cyclopleged with cycloplegic drops and will be refracted to obtain a cyclopleged refraction. This will determine his refractive error.
  Interventions: Device: Spot photoscreener; Procedure: Ophthalmologic evaluation; Procedure: Cyclopleged refraction

INTERVENTIONS:
Device: Spot photoscreener — Screening of vision problem through an automated device
Procedure: Ophthalmologic evaluation — Screening of vision problem through an ophthalmologic evaluation
Procedure: Cyclopleged refraction — Screening of refractive problems through a cyclopleged optometric refraction

SUMMARY:
Screening of haitian children between the ages of 3 and 6 years old for amblyogenic risk factors with the use of the Spot photoscreener. The photoscreener results will be compared to the complete ophthalmologic evaluation. Primarily, this will allow evaluation of the performance of the spot photoscreener in the haitian children population. Secondarily, this study will gather epidemiological information on vision problems in the haitian children population.

DETAILED DESCRIPTION:
Screening of haitian children between the ages of 3 and 6 years old for amblyogenic risk factors with the use of the Spot photoscreener before and after cycloplegia. The photoscreener results will be compared to the complete ophthalmologic evaluation. The ophthalmologic evaluation includes visual acuity, ocular alignment, slit lamp evaluation, cycloplegic refraction and dilated fundus evaluation. First of all, this will allow evaluation of the performance of the spot photoscreener in the haitian children population. Second of all, this study will gather epidemiological information on vision problems in the haitian children population.

ELIGIBILITY:
Inclusion Criteria:

* Haitian children aged 3-6 years of age
* Signed consent form from a legal guardian

Exclusion Criteria:

* Previous vision problem diagnostic
* Unsigned consent form

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Haitian children aged 3-6 years of age in Limbé, plaine du Nord and Port-au-Prince
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-01; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Number of patients presenting significant ophthalmologic pathologies in an haitian pediatric population | 7 days
  The epidemiology of vision problems will be evaluated in a sample of haitian children. The ophthalmologic exam will be considered abnormal if it denotes a significant ophthalmologic pathology. A significant ophthalmologic pathology is defined as a significant refractive error, a significant strabismus or a significant media opacity according to the 2013 American Association for Pediatric Ophthalmology and Strabismus (AAPOS) Guidelines for automated preschool vision screening. An ophthalmologic pathology is also considered significant in cases of severe ophthalmologic pathologies (xerophthalmia, trachoma, cataract >1mm, glaucoma, retinopathy of prematurity, retinoblastoma).

SECONDARY OUTCOMES:
Performance of the Spot photoscreeners in comparison with the ophthalmologic exam to denote significant ophthalmologic pathologies according to the 2013 AAPOS guidelines in an haitian pediatric population | 7 days
  Sensitivity, specificity, positive predictive value and negative predictive value of the abnormal automated vision screening with the photoscreener in comparison of the abnormal screening of the ophthalmologic exam using the criteria of the AAPOS guidelines (gold standard). A significant ophthalmologic pathology is defined as a significant refractive error, a significant strabismus or a significant media opacity according to the 2013 American Association for Pediatric Ophthalmology and Strabismus (AAPOS). The results of the test, being normal vs abnormal, will be compared.
Performance of the Spot photoscreeners in comparison with the ophthalmologic exam to denote severe ophthalmologic pathologies that are not described in the 2013 AAPOS guidelines in an haitian pediatric population | 7 days
  Sensitivity, specificity, positive predictive value and negative predictive value of the abnormal automated vision screening with the photoscreener in comparison of the abnormal screening of the ophthalmologic exam for all other severe ophthalmologic pathologies not described in the AAPOS guidelines (gold standard). An ophthalmologic pathology is also considered significant in cases of severe ophthalmologic pathologies (xerophthalmia, trachoma, cataract >1mm, glaucoma, retinopathy of prematurity, retinoblastoma). The results of the test, being normal vs abnormal, will be compared.
Performance of the Spot photoscreeners in comparison with the cyclopleged optometric exam in an haitian pediatric population | 7 days
  Sensitivity, specificity of the refractive errors measured with the photoscreener compared to the refractive errors measured by the cyclopleged optometric exam (gold standard). The values of the refraction, in dioptries, will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Antoine Sylvestre-Bouchard, Principal Investigator — Université de Montréal; Patrick Hamel, MD, FRCS, Study Chair — Université de Montréal; Christelle Doyon, MD, Study Director — Université de Montréal
Locations (3):
- Haiti (3):
  - École Adventiste de Limbé, Lenbe
  - ClinicA, Pétionville
  - École Saint-Dominique de Plaine du nord, Plaine du Nord

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maida JM, Mathers K, Alley CL. Pediatric ophthalmology in the developing world. Curr Opin Ophthalmol. 2008 Sep;19(5):403-8. doi: 10.1097/ICU.0b013e328309f180. PMID 18772673
- [Background] Resnikoff S, Pascolini D, Mariotti SP, Pokharel GP. Global magnitude of visual impairment caused by uncorrected refractive errors in 2004. Bull World Health Organ. 2008 Jan;86(1):63-70. doi: 10.2471/blt.07.041210. PMID 18235892
- [Background] Braverman R. Diagnosis and treatment of refractive errors in the pediatric population. Curr Opin Ophthalmol. 2007 Sep;18(5):379-83. doi: 10.1097/ICU.0b013e328244dfed. PMID 17700230
- [Background] Mathers M, Keyes M, Wright M. A review of the evidence on the effectiveness of children's vision screening. Child Care Health Dev. 2010 Nov;36(6):756-80. doi: 10.1111/j.1365-2214.2010.01109.x. PMID 20645997
- [Background] Krumholtz I. Results from a pediatric vision screening and its ability to predict academic performance. Optometry. 2000 Jul;71(7):426-30. PMID 15326895
- [Background] Atkinson J, Anker S, Nardini M, Braddick O, Hughes C, Rae S, Wattam-Bell J, Atkinson S. Infant vision screening predicts failures on motor and cognitive tests up to school age. Strabismus. 2002 Sep;10(3):187-98. doi: 10.1076/stra.10.3.187.8125. PMID 12461713
- [Background] Williams WR, Latif AH, Hannington L, Watkins DR. Hyperopia and educational attainment in a primary school cohort. Arch Dis Child. 2005 Feb;90(2):150-3. doi: 10.1136/adc.2003.046755. PMID 15665167
- [Background] Roch-Levecq AC, Brody BL, Thomas RG, Brown SI. Ametropia, preschoolers' cognitive abilities, and effects of spectacle correction. Arch Ophthalmol. 2008 Feb;126(2):252-8; quiz 161. doi: 10.1001/archophthalmol.2007.36. PMID 18268218
- [Background] Lennerstrand G, Jakobsson P, Kvarnstrom G. Screening for ocular dysfunction in children: approaching a common program. Acta Ophthalmol Scand Suppl. 1995;(214):26-38; discussion 39-40. doi: 10.1111/j.1600-0420.1995.tb00585.x. PMID 8574881
- [Background] Weinstock VM, Weinstock DJ, Kraft SP. Screening for childhood strabismus by primary care physicians. Can Fam Physician. 1998 Feb;44:337-43. PMID 9512837
- [Background] Williams C, Harrad RA, Harvey I, Sparrow JM; ALSPAC Study Team. Screening for amblyopia in preschool children: results of a population-based, randomised controlled trial. ALSPAC Study Team. Avon Longitudinal Study of Pregnancy and Childhood. Ophthalmic Epidemiol. 2001 Dec;8(5):279-95. doi: 10.1080/09286586.2001.11644257. PMID 11922382
- [Background] Williams C, Northstone K, Harrad RA, Sparrow JM, Harvey I; ALSPAC Study Team. Amblyopia treatment outcomes after screening before or at age 3 years: follow up from randomised trial. BMJ. 2002 Jun 29;324(7353):1549. doi: 10.1136/bmj.324.7353.1549. PMID 12089090
- [Background] Fathy VC, Elton PJ. Orthoptic screening for three- and four-year-olds. Public Health. 1993 Jan;107(1):19-23. doi: 10.1016/s0033-3506(05)80488-3. No abstract available. PMID 8475239
- [Background] Atkinson J, Braddick O, Robier B, Anker S, Ehrlich D, King J, Watson P, Moore A. Two infant vision screening programmes: prediction and prevention of strabismus and amblyopia from photo- and videorefractive screening. Eye (Lond). 1996;10 ( Pt 2):189-98. doi: 10.1038/eye.1996.46. PMID 8776448
- [Background] Atkinson J, Braddick O, Nardini M, Anker S. Infant hyperopia: detection, distribution, changes and correlates-outcomes from the cambridge infant screening programs. Optom Vis Sci. 2007 Feb;84(2):84-96. doi: 10.1097/OPX.0b013e318031b69a. PMID 17299337
- [Background] Kvarnstrom G, Jakobsson P, Lennerstrand G. Screening for visual and ocular disorders in children, evaluation of the system in Sweden. Acta Paediatr. 1998 Nov;87(11):1173-9. doi: 10.1080/080352598750031176. PMID 9846920
- [Background] Kvarnstrom G, Jakobsson P, Lennerstrand G. Visual screening of Swedish children: an ophthalmological evaluation. Acta Ophthalmol Scand. 2001 Jun;79(3):240-4. doi: 10.1034/j.1600-0420.2001.790306.x. PMID 11401631
- [Background] Eibschitz-Tsimhoni M, Friedman T, Naor J, Eibschitz N, Friedman Z. Early screening for amblyogenic risk factors lowers the prevalence and severity of amblyopia. J AAPOS. 2000 Aug;4(4):194-9. doi: 10.1067/mpa.2000.105274. PMID 10951293
- [Background] Jewell G, Reeves B, Saffin K, Crofts B. The effectiveness of vision screening by school nurses in secondary school. Arch Dis Child. 1994 Jan;70(1):14-8. doi: 10.1136/adc.70.1.14. PMID 8110000
- [Background] Cummings GE. Vision screening in junior schools. Public Health. 1996 Nov;110(6):369-72. doi: 10.1016/s0033-3506(96)80010-2. PMID 8979754
- [Background] Williams C, Northstone K, Harrad RA, Sparrow JM, Harvey I; ALSPAC Study Team. Amblyopia treatment outcomes after preschool screening v school entry screening: observational data from a prospective cohort study. Br J Ophthalmol. 2003 Aug;87(8):988-93. doi: 10.1136/bjo.87.8.988. PMID 12881342
- [Background] Snowdon SK, Stewart-Brown SL. Preschool vision screening. Health Technol Assess. 1997;1(8):i-iv, 1-83. PMID 9483159
- [Background] Shamanna BR, Dandona L, Rao GN. Economic burden of blindness in India. Indian J Ophthalmol. 1998 Sep;46(3):169-72. PMID 10085631
- [Background] Latorre-Arteaga S, Gil-Gonzalez D, Enciso O, Phelan A, Garcia-Munoz A, Kohler J. Reducing visual deficits caused by refractive errors in school and preschool children: results of a pilot school program in the Andean region of Apurimac, Peru. Glob Health Action. 2014 Feb 13;7:22656. doi: 10.3402/gha.v7.22656. eCollection 2014. PMID 24560253
- [Background] Kedir J, Girma A. Prevalence of refractive error and visual impairment among rural school-age children of Goro District, Gurage Zone, Ethiopia. Ethiop J Health Sci. 2014 Oct;24(4):353-8. doi: 10.4314/ejhs.v24i4.11. PMID 25489200
- [Background] Sommer A, Toureau S, Cornet P, Midy C, Pettiss ST. Xerophthalmia and anterior segment blindness. Am J Ophthalmol. 1976 Sep;82(3):439-46. doi: 10.1016/0002-9394(76)90492-x. PMID 961794
- [Background] Duong HV, Westfield KC, Jones LS, Mitchell J, Carr T. A survey of ocular diseases in an isolated rural Haitian community: a retrospective evaluation. J Natl Med Assoc. 2012 Nov-Dec;104(11-12):536-43. doi: 10.1016/s0027-9684(15)30220-0. PMID 23560356
- [Background] Courtright P, Hutchinson AK, Lewallen S. Visual impairment in children in middle- and lower-income countries. Arch Dis Child. 2011 Dec;96(12):1129-34. doi: 10.1136/archdischild-2011-300093. Epub 2011 Aug 24. PMID 21868404
- [Background] Kirk S, Armitage MD, Dunn S, Arnold RW. Calibration and validation of the 2WIN photoscreener compared to the PlusoptiX S12 and the SPOT. J Pediatr Ophthalmol Strabismus. 2014 Sep-Oct;51(5):289-92. doi: 10.3928/01913913-20140701-01. Epub 2014 Jul 8. PMID 25000209
- [Background] Silbert DI, Matta NS. Performance of the Spot vision screener for the detection of amblyopia risk factors in children. J AAPOS. 2014 Apr;18(2):169-72. doi: 10.1016/j.jaapos.2013.11.019. PMID 24698615
- [Background] Arnold RW, Armitage MD. Performance of four new photoscreeners on pediatric patients with high risk amblyopia. J Pediatr Ophthalmol Strabismus. 2014 Jan-Feb;51(1):46-52. doi: 10.3928/01913913-20131223-02. Epub 2014 Jan 3. PMID 24369683
- [Background] Sharma A, Congdon N, Patel M, Gilbert C. School-based approaches to the correction of refractive error in children. Surv Ophthalmol. 2012 May-Jun;57(3):272-83. doi: 10.1016/j.survophthal.2011.11.002. Epub 2012 Mar 6. PMID 22398336
- [Background] Donahue SP, Arthur B, Neely DE, Arnold RW, Silbert D, Ruben JB; POS Vision Screening Committee. Guidelines for automated preschool vision screening: a 10-year, evidence-based update. J AAPOS. 2013 Feb;17(1):4-8. doi: 10.1016/j.jaapos.2012.09.012. Epub 2013 Jan 27. PMID 23360915
- [Background] US Preventive Services Task Force. Vision screening for children 1 to 5 years of age: US Preventive Services Task Force Recommendation statement. Pediatrics. 2011 Feb;127(2):340-6. doi: 10.1542/peds.2010-3177. Epub 2011 Jan 31. PMID 21282267
- [Background] Committee on Practice and Ambulatory Medicine and Section on Ophthalmology; American Academy of Pediatrics. Use of photoscreening for children's vision screening. Pediatrics. 2002 Mar;109(3):524-5. doi: 10.1542/peds.109.3.524. PMID 11875154
- [Background] Arnold RW, Clausen M, Ryan H, Leman RE, Armitage D. Predictive value of inexpensive digital eye and vision photoscreening: "PPV of ABCD". Binocul Vis Strabismus Q. 2007;22(3):148-52. PMID 17983349